CLINICAL TRIAL: NCT05264896
Title: Perioperative FLOT Versus Adjuvant XELOX for Locally Advanced Gastric Cancer - a Randomized Controlled Study
Brief Title: Perioperative FLOT vs Adjuvant XELOX for CA Stomach
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2020.500
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Cancer of Stomach, Adenocarcinoma
Keywords: Gastric cancer; Cancer of esophagogastric junction; Chemotherapy; FLOT
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; XELOX

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FLOT (Experimental): Patients randomized to the FLOT arm would receive perioperative FLOT
  Regimen:
  * Docetaxel 50mg/m2, d1
  * 5-FU 2600 mg/m², d1
  * Leucovorin 200 mg/m², d1
  * Oxaliplatin 85 mg/m², d1
  * Every two weeks 4 cycles pre-op and 4 cycles post-op
  Granulocyte colony stimulating factor (GCSF) at 30 mu s.c. daily from Day 4 to Day 7 is recommended.
  Two weeks after completion of the 4 cycles of pre-op chemotherapy, reassessment endoscopy and CT scan would be performed. Surgery would be performed 4 weeks after pre-op chemotherapy if no distant metastasis was found on CT scan.
  Post-op adjuvant FLOT (x 4 cycles) will be started within 10 weeks after surgery.
  Interventions: Drug: 5-FU, Leucovorin, Oxaliplatin, Docetaxel
- XELOX (Active Comparator): Patients randomized to adjuvant XELOX arm would receive chemotherapy after surgery.
  * Capecitabine - 1,000 mg/m² twice daily.
  * Oxaliplatin - IV infusion, 130mg/m²
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: 5-FU, Leucovorin, Oxaliplatin, Docetaxel — FLOT 4 cycles pre and post radical gastrectomy
  Arms: FLOT
Drug: XELOX — XELOX 8 cycles post radical gastrectomy
  Arms: XELOX

SUMMARY:
This is a single centre randomised controlled trial, comparing perioperative FLOT versus adjuvant XELOX for locally advanced gastric and esophagogastric junction cancers. Patients with operable clinical T3 or above and N1 or above gastric and esophagastric junction cancer would be recruited. Participants would be randomised to perioperative FLOT versus adjuvant XELOX with curative radical gastrectomy. Primary outcome would be 3 year Disease Free Survival. It was calculated that 110 patients would be required to demonstrate the study hypothesis.

DETAILED DESCRIPTION:
The use of perioperative chemotherapy / chemoradiation for locally advanced cancer of the stomach and esophagogastric junction has been advocated in the past 2 decades. Randomized studies from Asia, Europe and the United States all demonstrated superior disease free survival with the use of perioperative therapy1-4. While radical gastrectomy plus D2 lymphadenectomy is the standard treatment in the treatment algorithm, the regimen of perioperative therapy has not been standardized. Earlier studies conducted in Europe and the United States using perioperative Epirubicin, Cisplatin, 5-FU (ECF) or postoperative chemoradiation were criticized owing to inadequate lymph node dissection. Adjuvant chemotherapy with either combination Capacitabine and Oxaliplatin or single agent S-1 has been proven in large prospective randomized studies in Asia, and these regimens are most commonly utilized currently.

Perioperative combination chemotherapeutic regimen using 5-FU, Leucovorin, Oxaliplatin and Docetaxel (FLOT) has been recently recommended in European countries. Initial phase II study demonstrated a dramatic improvement in complete tumor response rate (TRG1a) at 20% compared with 6% for ECF5. Results from a phase III randomized study showed superior overall survival using FLOT when compared with ECF (Median survival ECX/ECF 35months, FLOT 50 months, p=0.012)6. Radical surgery has been standardized in these recent studies. Another randomized study from Asia reported superior disease free survival when Docetaxel, Oxaliplatin and S-1 were used as pre-operative chemotherapy plus adjuvant S-1 monotherapy compared with S-1 monotherapy alone. (NCT01515748, abstract at ESMO 2019, Spain)

The main advantages of perioperative chemotherapy include downstaging of the tumor allowing easier and more complete surgical resection. The compliance rate to preoperative chemotherapy is also generally higher than postoperative therapy. Some may propose that it may also aid in selecting appropriate cases for radical surgery, thus avoiding unnecessary surgery in those who progress quickly. However, the potential drawback of such treatment regimen includes higher risk of surgery after chemotherapy and potential delay of curative surgery.

There is currently lack of prospective comparative data between adjuvant XELOX and perioperative FLOT. Our institution decided to conduct the current study to compare the survival outcomes of locally advanced cancer of stomach and esophagogastric junction after perioperative FLOT or adjuvant XELOX plus radical surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced adenocarcinoma of stomach or esophagogastric junction (Siewert type II and III), defined by clinical stage ≥T3 and/or ≥N1, in the absence of distant metastasis
2. Surgically resectable disease based on clinical staging
3. No previous gastrectomy or chemotherapy
4. Age 18 or above but less than 80, and
5. ECOG ≤2
6. Hemoglobin >/= 8.0 g/dL
7. Neutrophils >/= 1.500/µl
8. Platelets ≥ 100.000/µl
9. Creatinine clearance ≥ 50 ml/min
10. Serum albumin >25 g/L

Exclusion criteria:

1. Distant metastases, direct tumor invasion to organs not resectable by surgery
2. Hypersensitivity or contraindication against Capacitabine, 5-FU, Leucovorin, Oxaliplatin, Docetaxel
3. Active CHD, Cardiomyopathy or cardiac insufficiency stage III-IV according to NYHA
4. Peripheral polyneuropathy ≥ NCI grade II
5. Severe liver dysfunction (i) ALT >3 x upper limit of normal, and/ or (ii) total bilirubin >1.5 x upper limit of normal (subjects with Gilbert Syndrome with total bilirubin level of >/= 3.0 x upper limit of normal)
6. Pregnancy or lactation
7. Malignant secondary disease, dated back <5 years (except in-situ carcinoma of cervix uteri, adequately treated skin basal cell carcinoma)
8. Serious uncontrolled infection or cocomitant severe medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3 year disease free survival | 3 years
  3 year disease free survival (%)

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival (%)
Adverse event of chemotherapy | 6 months
  Adverse event of chemotherapy (%)
Adverse event of surgery | 30 days
  Adverse event of surgery (%)
Rate of completion of all cycles of chemotherapy | 1 year
  Completion rate of all cycles of chemo (%)
Postoperative hospital stay | 3 months
  Postoperative hospital stay (days)
Recurrence | 5 years
  Rate of Locoregional or distant recurrence
Pathology - tumor regression grade | 30 days
  Pathology - Tumor Regression Grade (Based on Becker's scale) TRG 1a was defined as complete tumor regression without residual tumor; TRG 1b was defined as <10% residual tumor per tumor bed, like a subtotal tumor regression. TGR 2 illustrated a partial tumor regression with 10-50% residual tumor and at the findings of >50% residual tumor cells with or without signs of treatment effect the tumor regression was classified as TRG 3

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No